CLINICAL TRIAL: NCT04886999
Title: An Exploratory, Double-blind, Randomised, Multicenter, Psychopharmacological Study in Adult Patients With Moderate to Severe Asthma to Compare Two Pressurised Metered-Dose Inhalers (pMDIs) on Patients' Perception of Asthma Symptoms
Brief Title: Study in Adult Patients With Moderate to Severe Asthma
Acronym: FEEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CLI-01535AA0-02; 2021-001449-11 (EudraCT Number)
Record Dates: First submitted 2021-04-27; First posted 2021-05-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Exploratory, double-blind, randomised, multicenter, 2x2 cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Exploratory, double-blind, randomised, multicenter, 2x2 cross-over study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaler A CHF1535 100/6 µg pMDI (Experimental): Active ingredient: Fixed combination of beclomethasone dipropionate 100 µg plus formoterol fumarate 6 µg.
  Excipients: HFA-134a, Ethanol anhydrous, Hydrochloric acid. Presentation: Canister containing 120 doses plus actuator.
  Interventions: Behavioral: Exploratory study on patient's perception of Asthma symptoms
- Inhaler B CHF1535 100/6 µg pMDI (Active Comparator): Active ingredient: Fixed combination of beclomethasone dipropionate 100 µg plus formoterol fumarate 6 µg.
  Excipients: HFA-134a, Ethanol anhydrous, Hydrochloric acid. Presentation: Canister containing 120 doses plus actuator
  Interventions: Behavioral: Exploratory study on patient's perception of Asthma symptoms

INTERVENTIONS:
Behavioral: Exploratory study on patient's perception of Asthma symptoms — To assess the perception of symptoms and the psychopharmacological aspects in patients with moderate to severe asthma comparing two inhalers of CHF1535 100/6 µg pMDI

SUMMARY:
The CLI-01535AA02-2 Study is an exploratory study designed to compare two pressurised metered Dose inhalers on subject's perception of asthma symptoms.

DETAILED DESCRIPTION:
Outpatients attending the hospital clinics/study centers will be recruited. Moderate to severe asthma adult subjects will be recruited. A total of 75 subjects will be enrolled. The whole study will last approximately 6 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject's and/or subject legal representative's written informed consent obtained prior to any study related procedure.
* Age: ≥18 and ≤75 years of age.
* Established diagnosis of permanent asthma for at least 6 months prior to screening/randomisation visit
* Subject on maintenance therapy treated by Foster® (CHF1535 100/6 µg pMDI) for at least 6 months prior to screening/randomisation visit
* Asthma Control Test (ACT) ≥ 20 at screening/randomisation visit.
* Subject must have a cooperative attitude and the ability to be trained to use correctly the diary and answer the Visual Analogue Scale (VAS)
* Subject willing and able to download the application on their personal electronic device to fill in the study e-diary.
* Female subject of non-childbearing potential defined as physiologically incapable of becoming pregnant or female subject + male Partner must be willing to use a highly effective birth control method from the signature of the informed consent and until Visit 4

Exclusion Criteria:

* Pregnant or lactating woman
* History of 'at risk' asthma
* Recent exacerbation
* Non-permanent asthma
* Asthma requiring more than 1 inhaler for maintenance treatment and more than 1 inhaler for reliever treatment.
* Asthma requiring use of biologics
* Respiratory disorders
* Lower tract respiratory infection
* Current smoker or ex-smoker with a smoking current use/history of ≥ 10 pack-years
* Cardiovascular diseases
* subject with historical or current evidence of uncontrolled concurrent disease such as but not limited to hyperthyroidism, diabetes mellitus or other endocrine disease; haematological disease; autoimmune disorders
* Alcohol/drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Summary measures (for questions with continuous outcome) to report patients' expectations of their symptoms change at Day 15 (Visit 2) | At Day 15 (Visit 2)
  Assessed by Visual Analogue Scale (VAS) that ranges from 0 to 100. When question refers to symptom improvement, higher score means better outcome. When question refers to symptoms worsening, higher score means worse outcome.
  Each question will be analysed separately.
Summary measures (for questions with continuous outcome) to report patients' expectations of their symptoms change at Day 29 (Visit 3) | At Day 29 (Visit 3)
  Assessed by Visual Analogue Scale (VAS) that ranges from 0 to 100. When question refers to symptom improvement, higher score means better outcome. When question refers to symptoms worsening, higher score means worse outcome.
  Each question will be analysed separately.
Summary measures (for questions with continuous outcome) to report patients' expectations of their symptoms change at Day 43 (Visit 4) | At Day 43 (Visit 4)
  Assessed by Visual Analogue Scale (VAS) that ranges from 0 to 100. When question refers to symptom improvement, higher score means better outcome. When question refers to symptoms worsening, higher score means worse outcome.
  Each question will be analysed separately.
Percentages of subjects (for questions with categorical outcome) to evaluate patients' preference of device at Day 43 (Visit 4) | At Day 43 (Visit 4)
  Questions covering patients' preference of device and outcome assessments will be reported on the ITT and PP set by treatment group. This analysis will be applied on questions not collected daily. Each question will be analysed separately.
Percentages of subjects (for questions with categorical outcome) to evaluate patients' perception of inhalers changes at Day 43 (Visit 4) | At Day 43 (Visit 4)
  Questions covering patients' preference of device and outcome assessments will be reported on the ITT and PP set by treatment group. This analysis will be applied on questions not collected daily. Each question will be analysed separately.
Change from baseline in average Visual Analogic Scale score of subjects' perceptions of asthma symptoms after 14 days of treatment | After 14 days of treatment
  Visual Analogue Scale (VAS) ranges from 0 to 100. When question refers to symptom improvement, higher score means better outcome. When question refers to symptoms worsening, higher score means worse outcome.
Change from baseline in average Visual Analogic Scale score of subjects' perceptions of asthma symptoms after the first 7 days of treatment | After the first 7 days of treatment
  Visual Analogue Scale (VAS) ranges from 0 to 100. When question refers to symptom improvement, higher score means better outcome. When question refers to symptoms worsening, higher score means worse outcome.
Change from baseline in rescue medication use | After 14 days of treatment
  To be summarised on the "Intention To Treat" set by treatment group by descriptive statistics. Baseline value is defined as the average value (puffs/day) collected during the baseline period.
Change from baseline in Asthma Quality of Life Questionnaire (AQLQ) score | After 14 days of treatment
  There are 32 questions in the AQLQ that are divided in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Answers are done on a 7-point scale (7 = not impaired at all - 1 = severely impaired), with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Event (TEAEs), adverse drug reactions (ADRs), severe ADRs, serious ADRs, serious TEAEs (Serious Adverse Events), non-serious TEAEs, severe TEAEs | From date of the first study drug intake unil date of study treatment, or date of death or up to 14 days after date of the last study drug intake, whichever came first
  Occurrence of Treatment Emergent Adverse Event (TEAEs), adverse drug reactions (ADRs), severe ADRs, serious ADRs, serious TEAEs (Serious Adverse Events), non-serious TEAEs, severe TEAEs, TEAEs leading to discontinuation from study treatment and TEAEs leading to death.
  Summarised on the safety set by treatment group as the number of subjects, percentage of subjects, and number of events. All adverse events starting on or after the time of first study drug intake will be classified as TEAE. Any adverse events started after the informed consent signature and before the time of first study drug intake will be classified as pre-treatment adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Topole, MD, Study Director — Chiesi Farmaceutici S.p.A.
Locations (10):
- Italy (10):
  - Chiesi 38011, Bari
  - Chiesi 38009, Battipaglia
  - Chiesi 38006, Cagliari
  - Chiesi 38010, Catanzaro
  - Chiesi 38003, Genova
  - Chiesi 38001, Milan
  - Chiesi 38005, Napoli
  - Chiesi 38004, Palermo
  - Chiesi 38002, Roma
  - Chiesi 38007, Sassari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2021-001449-11/results